CLINICAL TRIAL: NCT05139238
Title: Oral Nifedipine Versus Intravenous Labetalol for Postpartum (PP) Hypertensive Emergency: A Randomized Clinical Trial (RCT)
Brief Title: Postpartum Hypertension Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Whitney Booker, Assistant Professor of Obstetrics and Gynecology, Columbia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AAAT5925
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-02

CONDITIONS: Postpartum Pregnancy-Induced Hypertension; Postpartum Preeclampsia; Pregnancy-Induced Hypertension in Postpartum; Hypertensive Emergency
Keywords: Hypertension; Hypertensive Emergency; Postpartum; Preeclampsia
MeSH Terms: conditions — Hypertensive Crisis; Hypertension; Pre-Eclampsia | interventions — Labetalol; Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Nifedipine (Active Comparator): Oral nifedipine: Once diagnosis of hypertensive emergency is confirmed on repeat blood pressure, patients randomized to oral nifedipine will receive 10mg initially, with repeated doses of 20mg every 20min, for up to a maximum of 5 doses or until the therapeutic blood pressure goal of <160 systolic and <105 diastolic is achieved. If the therapeutic goal is not achieved after 5 doses, crossover to the alternative study medication will occur.
  Interventions: Drug: Nifedipine
- Intravenous labetalol (Active Comparator): Intravenous Labetalol: Patients randomized to IV labetalol will receive 20mg initially, followed by escalating doses of 40mg, 80mg, 80mg, then 80mg every 20 minutes until the therapeutic goal is achieved, for a maximum of 5 doses. If the therapeutic goal is not achieved after 5 doses, crossover to the alternative study medication will occur.
  Interventions: Drug: Labetalol

INTERVENTIONS:
Drug: Labetalol — Intravenous labetalol, a short acting ant-hypertensive
  Arms: Intravenous labetalol
Drug: Nifedipine — Oral nifedipine, a short acting ant-hypertensive
  Other Names: Oral Procardia
  Arms: Oral Nifedipine

SUMMARY:
The purpose of this study is to assess which blood pressure medication (intravenous labetalol or oral nifedipine) works better in treating severely elevated blood pressure in women who have just delivered a baby.

DETAILED DESCRIPTION:
Hypertensive emergencies cause significant maternal morbidity and mortality in the postpartum period. In order to reduced these risks, the recommendation is to treat women with severe range blood pressure with either intravenous labetalol or oral nifedipine; it is unclear which medication is superior. The objective of this study is to prospectively enroll women who have hypertensive emergencies in the postpartum period; women will be randomized in a 1:1 fashion and treated with one of the two antihypertensives to see which one works better.

ELIGIBILITY:
Inclusion criteria

* Patients admitted to labor and delivery (L&D) with blood pressure (BP) in severe range, defined as a systolic ≥160 mm Hg and/or diastolic ≥110 mm Hg
* Postpartum, immediately to 6 weeks postpartum
* With a prior diagnosis of chronic hypertension (not on medication) or hypertensive disorder of pregnancy

Exclusion criteria

* They may not have previously had exposure to either study medication within the previous 24-hour period.
* Patients with a known atrial-ventricular heart block or moderate to severe bronchial asthma will be excluded, or other contraindication to receiving either study medication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Average Time to Initial Blood Pressure Control (minutes) | Up to 48 hours
  The primary outcome will be time (minutes) interval required to achieve the therapeutic BP goal of <160 mmHg systolic and <110 mmHg diastolic.

SECONDARY OUTCOMES:
Average Number of Recurrence of Severe Blood Pressure | Up to 48 hours
  The number of times a patient has recurrence of severe hypertensive necessitating treatment with an antihypertensive.
Total Number of Participants Who Need for Second Antihypertensive Agent | Up to 48 hours
  The need to use a second (alternative) antihypertensive medication.

CONTACTS AND LOCATIONS:
Overall Officials: Whitney A. Booker, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided